CLINICAL TRIAL: NCT05455411
Title: A Predict-to-Prescribe Approach to Social Communication Treatment in Chinese Preschool Children With Autism Spectrum Disorder
Brief Title: Parent-implemented Social Communication Treatment in Preschool Children With Autism Spectrum Disorder
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Patrick C. M. Wong, Stanley Ho Professor of Cognitive Neuroscience; Director of Brain and Mind Institute, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CRFASD-22
Record Dates: First submitted 2022-06-29; First posted 2022-07-13 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Autism Spectrum Disorder; Autism; Social Communication; Speech Therapy; Parenting
Keywords: Autism Spectrum Disorder; Parent-implemented Intervention; Social Communication
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder; Communication; Communication Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group-based Parent-implemented Social Communication Training (Experimental): A group-based parent-implemented social communication treatment program for up to 8 parents of children with autism spectrum disorder
  Interventions: Behavioral: Group-based Parent-implemented Training
- Individual-based Parent-implemented Social Communication Training (Active Comparator): An individual-based parent-implemented social communication treatment program for a parent of a child with autism spectrum disorder
  Interventions: Behavioral: Individual-based Parent-implemented Training

INTERVENTIONS:
Behavioral: Group-based Parent-implemented Training — A group-based social communication training for parents of preschoolers with autism spectrum disorder will be taught by a speech therapist online (approximately 25 hours distributed over 6 months), with up to 8 parents in a group.
  Arms: Group-based Parent-implemented Social Communication Training
Behavioral: Individual-based Parent-implemented Training — An individual-based social communication training for parents of preschoolers with autism spectrum disorder will be taught by a speech therapist online in a one-on-one format (approximately 25 hours distributed over 6 months).
  Arms: Individual-based Parent-implemented Social Communication Training

SUMMARY:
An accumulation of research evidence has pointed to parent-implemented communication treatment as effective in reducing the severity of social communication deficits in preschool children with ASD. Despite even high-quality evidence, real-world translation to clinical practice remains challenging, especially for children from lower-income families, for two reasons. First, the treatment outcome is highly variable despite study-level efficacy data, most likely due to unique child and parent factors that make treatment response uneven across individual children. Second, the cost of intervention with the largest effect sizes remains high due to its one-on-one format.

With the overarching goal to reduce cost and to increase treatment effectiveness at the individual-child level, this project will conduct a randomized controlled trial (RCT) to compare the effectiveness of two options for intervention to address two specific objectives. The investigators will first ascertain whether parent-implemented communication treatment taught by a speech therapist in an Individual (one-on-one) format is more effective than treatment taught in a Group format (up to 8 families learning together) at the study level. The Individual format is at least 4 times more expensive than the Group format; its relative treatment effect must be empirically ascertained to justify its cost. The investigators will then evaluate what combinations of parent and child behavioral and neural factors determine which format of intervention is likely to be more effective at the individual-child level. It is likely that not all families require the more costly Individual format of intervention. Machine-learning analytics with cross-validation will be used in constructing predictive models of treatment response, which will increase the likelihood of these models being generalizable to new patients.

This study will be among the first examples of fulfilling the promise of Precision Medicine in providing guidance to patients and families with developmental disorders not about whether to receive intervention but which option for intervention to receive in the context of multiple options. This predict-to-prescribe approach of ASD intervention will likely lead to a paradigm shift in clinical practice and ultimately result in lowering the overall cost and increasing the effectiveness of intervention for children with ASD as individuals.

DETAILED DESCRIPTION:
BACKGROUND:

For parents of children with Autism Spectrum Disorder (ASD), the primary concern is to minimize the impact of the disorder, likely through evidence-based intervention. The secondary concern is whether any intervention prescribed is affordable and the logistics of completion feasible. This project will obtain evidence for ASD intervention options that have different costs and intervention delivery formats (individual vs. group) to evaluate whether a more costly option is more effective at the study level. The investigators will then develop a predict-to-prescribe approach that informs parents which intervention option would likely be most cost-effective in light of each family's unique characteristics (i.e., effectiveness at the individual-child level). [We use the term "parents" to mean caregivers throughout this protocol.]

ASD affects 14 per 10,000 (0.14%) children in Hong Kong and 39.23 per 10,000 in Mainland China. Social communication is a deficit domain of ASD, and about 29% of preschoolers with ASD have severe verbal deficits. Intervention through pharmaceutical means remains elusive, leaving behavioral interventions the most realistic and immediate avenue of treatment. This project will focus on enhancing the cost-effectiveness of behavioral intervention that targets language and communication. The investigators will do so in the context of precision medicine, in which the investigators aim to identify the most cost-effective intervention for the individual child with ASD.

AIM OF STUDY:

Objective 1: The investigators will first ascertain whether parent-implemented communication treatment taught by a speech therapist in an Individual (one-on-one) format is more effective than treatment taught in a Group format (up to 8 families learning together) at the study level.

Objective 2: The investigators will examine pre-treatment child and parent variables simultaneously and construct predictive models of response to the two treatment options (group, less costly vs. individual, more costly) at the individual-child level. Both neural and non-neural variables will be examined to increase the precision of prediction.

HYPOTHESIS:

By the investigators' estimate, even after the number of contact hours is controlled, the group format is at least 4 times cheaper than the one-on-one format. Individual sessions allow for individualization, clearer explanation and modeling of the strategies, as well as some clinician-to-child stimulations that cannot be achieved by lectures. Though it may seem obvious that this individual format must produce better results, it is possible that the group format may be more effective due to better social support offered by peers.

ELIGIBILITY:
Inclusion Criteria:

* Have a confirmed diagnosis of autism spectrum disorder or was evaluated to have elevated likelihood ("at-risk" or "suspected") by a Clinical Psychologist, Psychiatrist or Pediatrician who recommended continuous surveillance.
* ADOS-2 score in the spectrum range (for Modules 1 & 2) or mild-to-moderate concern range (for Toddler Module)

Exclusion Criteria:

* Mullen Scale of Early Learning non-verbal age at or less than 12 months
* Parent who has severe psychological or neurological conditions prohibiting them from conducting the treatment program at home (restricted to only the parent in the program)
* Children with any other severe developmental problems beyond autism spectrum disorder

Ages: 18 Months to 60 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 112 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Social Affect at 12 months | Baseline and at 12 months after the beginning of treatment
  Comparing the pre- and post-treatment social affect measured by the Social Affect subscore of Autism Diagnostic Observation Schedule™, Second Edition (ADOS-2) between groups.
  The Social Affect subscore of ADOS-2 ranges from 0 to 20; the higher ADOS-2 scores mean a worse outcome.

SECONDARY OUTCOMES:
Change from Baseline Number of Parent-child Turn-taking at 6 months and 12 months | Baseline, at 6 months and at 12 months after the beginning of treatment
  Comparing the pre- and post-treatment number of parent-child turn-taking between groups.
  A parent-child interaction video will be taken; the number of turn-taking will be counted. The greater number of the mentioned language and communication features mean a better outcome.
Change from Baseline Mean Length of Utterance at 6 months and 12 months | Baseline, at 6 months and at 12 months after the beginning of treatment
  Comparing the pre- and post-treatment mean length of utterance between groups.
  A parent-child interaction video will be taken; speech of children will be transcribed. The length of utterance will be assessed and the mean length of utterance will be calculated. The longer mean length of utterance mean a better outcome.
Change from Baseline Number of Nouns and Verbs at 6 months and 12 months | Baseline, at 6 months and at 12 months after the beginning of treatment
  Comparing the pre- and post-treatment number of nouns and verbs between groups.
  A parent-child interaction video will be taken; speech of children will be transcribed. The number of nouns and verbs will be counted. The greater number of nouns and verbs means a better outcome.
Change from Baseline Prosody in terms of loudness variation at 6 months and 12 months | Baseline, at 6 months and at 12 months after the beginning of treatment
  Comparing the pre- and post-treatment loudness variation between groups.
  A parent-child interaction video will be taken. Audio with the speech of children will be extracted. Loudness of the audio will be assessed with Praat, an acoustic analysis software. The reduction of the loudness variation means a better outcome.
Change from Baseline Prosody in terms of fundamental frequency at 6 months and 12 months | Baseline, at 6 months and at 12 months after the beginning of treatment
  Comparing the pre- and post-treatment fundamental frequency between groups.
  A parent-child interaction video will be taken. Audio with the speech of children will be extracted. The fundamental frequency of the audio will be assessed with Praat, an acoustic analysis software. The reduction of fundamental frequency means a better outcome.

CONTACTS AND LOCATIONS:
Locations (2):
- Hong Kong (2):
  - The Chinese University of Hong Kong, Shatin
  - Castle Peak Hospital, Tuenmen

IPD SHARING:
Plan to Share IPD: No